CLINICAL TRIAL: NCT06709274
Title: Minimal Residual Disease (MRD)-Guided Adjuvant Therapy in Stage I Non-Small Cell Lung Cancer: A Prospective, Multicenter, Randomized Controlled Study
Brief Title: Minimal Residual Disease Guiding Adjuvant Therapy in Stage I NSCLC
Acronym: MOTION-NSCLC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: Nanjing Geneseeq Technology Inc. (Industry)
Responsible Party: Principal Investigator, Xue-Ning Yang, Principal Investigator, Guangdong Association of Clinical Trials
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG2301
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; alectinib; toripalimab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MRD-guided management (Experimental): Patients who are MRD-positive after surgery in the MRD-guided management group receive adjuvant therapy. Patients who are MRD-negative in the MRD-guided management group are monitored through observation.
  Interventions: Drug: Osimertinib; Drug: Alectinib; Drug: TORIPALIMAB INJECTION (JS001 ) combine with chemotherapy
- Standard of care (No Intervention): Adjuvant therapy is not recommended. However, if the physician and patient decide on adjuvant therapy, the treatment regimen and cycle must be documented. Researchers are strongly advised to follow the medication guidelines laid out in the Chinese Society of Clinical Oncology (CSCO) Clinical Practice Guidelines.

INTERVENTIONS:
Drug: Osimertinib — 80mg daily, for EGFR-positive patients
  Arms: MRD-guided management
Drug: Alectinib — 600mg BID, for ALK-rearranged patients
  Arms: MRD-guided management
Drug: TORIPALIMAB INJECTION (JS001 ) combine with chemotherapy — Toripalimab 240mg + Platinum-based chemotherapy (Q3W for 4 cycles), followed by Toripalimab maintenance therapy (240mg Q3W for one year), for EGFR/ALK wildtype patients
  Arms: MRD-guided management

SUMMARY:
This investigator-initiated study aims to evaluate the effectiveness of minimal residual disease (MRD) as a biomarker for guiding adjuvant therapy decisions in patients with Stage I non-small-cell lung cancer (NSCLC). The study will compare outcomes between an MRD-guided management group and a standard-of-care group, focusing on whether the use of MRD information can improve the 3-year disease-free survival rate compared to existing treatment protocols. Participants in the MRD-guided management group will receive targeted therapy, immunotherapy, or observation based on their postoperative MRD status, while those in the standard-of-care group will receive treatments or observation according to current clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Non-small cell lung cancer (NSCLC) confirmed by histological and/or cytological examination. Invasive subtypes are required for adenocarcinomas.
2. Stage IA or IB after surgery based on pathological TNM8 staging criteria established by the International Union Against Cancer/American Joint Committee on Cancer (8th Edition).
3. Completely surgical resection (R0) of the primary NSCLC via lobectomy, segmentectomy, or sleeve lobectomy. The gross tumor must be entirely removed, and all surgical margins of the excised tumor must be negative.
4. Complete recovery from surgery with no evidence of disease progression within 2 weeks prior to the first treatment decision.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
6. Minimum life expectancy of ≥12 weeks.
7. Demonstrate adequate organ function, including:

   Hematological parameters:
   * Absolute neutrophil count ≥1.5×10^9/L
   * Platelet count ≥100×10^9/L
   * Hemoglobin ≥90 g/L

   Liver function:
   * ALT ≤2.5× upper limit of normal (ULN)
   * AST ≤2.5×ULN
   * Total Bilirubin (TBL) ≤1.5×ULN Renal function: Creatinine level ≤1.25×ULN, or creatinine clearance ≥60 mL/min (measured or calculated using the Cockcroft-Gault formula).
8. Male or female, age between 18 and 75 years.
9. Written informed consent must be obtained from the subject or their legal representative.
10. Participants regardless of sex must agree to use effective contraception during the study period and for 3 months following treatment completion.
11. Willingness and ability to comply with visit schedules, treatment plans, and laboratory assessments.

Exclusion Criteria:

1. Histopathologically confirmed small cell carcinoma components.
2. Presence of multiple pulmonary nodules.
3. Incomplete resections (R1/R2) or resections via bilateral lobectomy, pneumonectomy, or wedge resection.
4. A history of any systemic anti-tumor treatment, including but not limited to surgery, neoadjuvant chemotherapy, radiotherapy, targeted therapy, or immunotherapy.
5. Significant allergies to any targeted drugs, immunotherapies, or chemotherapy agents used in the study.
6. Previous use of any traditional Chinese medicine with anti-tumor properties, or use of such medicine within 2 weeks prior to surgery.
7. History of other malignancies within the past 5 years, with the exception of the following:

   * Other malignancies fully cured by surgery with a disease-free survival of more than 10 years
   * Curable basal cell carcinoma of the skin
   * Bladder carcinoma in situ
   * Cervical carcinoma in situ
8. History of interstitial lung disease, drug-induced interstitial lung disease, radiation-induced pneumonia requiring steroid treatment, or any evidence of clinically active interstitial lung disease.
9. Active hepatitis B, defined as HBsAg positive with an HBV-DNA copy number exceeding the ULN established by the study center, accompanied by abnormal liver function, or requiring treatment as evaluated by the investigator.
10. Presence of any unstable systemic disease, including but not limited to active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the past 3 months, serious arrhythmias that requires medication, liver disease, kidney disease, or metabolic disorders.
11. Evidence of any other diseases, neurological or metabolic disorders, or physical exam or laboratory findings that may suggest contraindications for the investigational drug, or a high risk for treatment-related complications.
12. Any of the following cardiac conditions:

    * Resting ECG QT interval (QTc) > 470 msec.
    * Significant abnormalities in rhythm, conduction, or morphology on resting ECG, including complete left bundle branch block, third-degree atrioventricular block, or second-degree atrioventricular block
    * Factors increasing the risk of QTc prolongation or arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, unexplained sudden death in a first-degree relative under the age of 40, or use of medications known to prolong QT interval.
13. Blood transfusion within 2 weeks prior to and during the surgery.
14. History of alcohol or drug abuse.
15. Pregnant or breastfeeding females.
16. Any other factors that the investigator deems may affect the progress of the study or compromise the trial data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
3-Year disease-free survival (DFS) Rate | 3 years post randomization
  The proportion of patients remain disease-free at the 3-year mark starting from the day of randomization

SECONDARY OUTCOMES:
5-Year disease-free survival (DFS) Rate | 5 years post randomization
  The proportion of patients remain disease-free at the 5-year mark starting from the day of randomization
5-Year overall survival (OS) rate | 5 years post randomization
  The proportion of patients remain alive at the 5-year mark starting from the day of randomization
Disease-free survival (DFS) | Up to 8 years post randomization
  Defined as the time from randomization to the first recorded instance of tumor recurrence or metastasis, whichever occurs first
Overall survival | Up to 8 years post randomization
  Defined as the time from the day of randomization to death from any cause
Quality of Life (QoL) Assessed using the EORTC QLQ-C30 (Version 3.0) | Up to 8 years post randomization
  Assessed using the EORTC QLQ-C30 (Version 3.0), developed by the European Organization for Research and Treatment of Cancer.
  EORTC QLQ-C30 (Version 3.0) is utilized to assess the overall quality of life in cancer patients. It measures a global health status/QoL scale, five functional scales, three symptom scales, and six single items. Each dimension is scored on a scale from 0 to 100, where a high score for the global health status/QoL represents a high QoL, a high score for a functional scale represents a high/healthy level of functioning, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of Life (QoL) Assessed using the EORTC QLQ-LC13 | Up to 8 years post randomization
  Assessed using the EORTC QLQ-LC13, developed by the European Organization for Research and Treatment of Cancer.
  EORTC QLQ-LC13 is a supplementary module focusing specifically on the quality of life of patients with lung cancer. It provides additional insights into symptoms and problems related to lung cancer and its treatment. Like the QLQ-C30, responses are measured on a scale from 0 to 100, where higher scores indicate greater severity of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long Wu, M.D., Principal Investigator — Guangdong Provincial People's Hospital; Xue-Ning Yang, M.D., Principal Investigator — Guangdong Provincial People's Hospital
Locations (15):
- China (15):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Guangdong Provincial People's Hostpital, Guangzhou, Guangdong
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Third People's Hospital of Chengdu, Chengdu, Sichuan